CLINICAL TRIAL: NCT04232839
Title: Formulation Selection and Subsequent Optimization of Two Different Oral Formulations of BI 894416 in Healthy Male Subjects (Open-label, Randomised, Single-dose Study in Two Parts; Trial Part 1: Five-period Crossover Design With an Additional Sixth Period in a Fixed Sequence; Trial Part 2: Three-period Crossover Followed by a Two-period Crossover Design)
Brief Title: A Study in Healthy Men to Find the Best Formulation of BI 894416 and to Test How This is Taken up in the Body
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to company decision.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1371-0022; 2019-003424-21 (EudraCT Number)
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- T3-R1-T1-T4-T2-T5 (sequence I+T5) (Experimental): Sequence I+T5, with treatments in the following order: T3-R1-T1-T4-T2-T5 with a washout period of at least 4 days between treatments. All test treatments (T1-T6) were one single dose of 62.5 milligram. R1 and T1-T4: taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. T5-T6: taken orally with 240 mL of water following a high-fat high-calorie breakfast.
  Reference (R1): 60 milligram (mg) (6 x 10 mg tablets) BI 894416 Reference Formulation, immediate release (IR) tablets.
  Test 1 (T1): 1 tablet BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR).
  Test 2 (T2): 1 tablet BI 894416 Formulation C2, ER tablet (slow release rate, SRR).
  Test 3 (T3): 1 capsule BI 894416 Formulation D2, ER capsule (FRR). Test 4 (T4): 1 capsule BI 894416 Formulation F2, ER capsule (SRR). Test 5 (T5): 1 tablet BI 894416 Formulation C2, ER tablet (SRR). Test 6 (T6): 1 capsule BI 894416 Formulation F2, ER capsule (SRR).
  Interventions: Drug: BI 894416 Reference Formulation; Drug: BI 894416 Formulation A2; Drug: BI 894416 Formulation C2; Drug: BI 894416 Formulation D2; Drug: BI 894416 Formulation F2
- T3-R1-T1-T4-T2-T6 (sequence I+T6) (Experimental): Sequence I+T6, with treatments in the following order: T3-R1-T1-T4-T2-T6 with a washout period of at least 4 days between treatments. All test treatments (T1-T6) were one single dose of 62.5 milligram. R1 and T1-T4: taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. T5-T6: taken orally with 240 mL of water following a high-fat high-calorie breakfast.
  Reference (R1): 60 milligram (mg) (6 x 10 mg tablets) BI 894416 Reference Formulation, immediate release (IR) tablets.
  Test 1 (T1): 1 tablet BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR).
  Test 2 (T2): 1 tablet BI 894416 Formulation C2, ER tablet (slow release rate, SRR).
  Test 3 (T3): 1 capsule BI 894416 Formulation D2, ER capsule (FRR). Test 4 (T4): 1 capsule BI 894416 Formulation F2, ER capsule (SRR). Test 5 (T5): 1 tablet BI 894416 Formulation C2, ER tablet (SRR). Test 6 (T6): 1 capsule BI 894416 Formulation F2, ER capsule (SRR).
  Interventions: Drug: BI 894416 Reference Formulation; Drug: BI 894416 Formulation A2; Drug: BI 894416 Formulation C2; Drug: BI 894416 Formulation D2; Drug: BI 894416 Formulation F2
- T2-T1-T3-R1-T4-T5 (sequence II+T5) (Experimental): Sequence II+T5, with treatments in the following order: T2-T1-T3-R1-T4-T5with a washout period of at least 4 days between treatments. All test treatments (T1-T6) were one single dose of 62.5 milligram. R1 and T1-T4: taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. T5-T6: taken orally with 240 mL of water following a high-fat high-calorie breakfast.
  Reference (R1): 60 milligram (mg) (6 x 10 mg tablets) BI 894416 Reference Formulation, immediate release (IR) tablets.
  Test 1 (T1): 1 tablet BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR).
  Test 2 (T2): 1 tablet BI 894416 Formulation C2, ER tablet (slow release rate, SRR).
  Test 3 (T3): 1 capsule BI 894416 Formulation D2, ER capsule (FRR). Test 4 (T4): 1 capsule BI 894416 Formulation F2, ER capsule (SRR). Test 5 (T5): 1 tablet BI 894416 Formulation C2, ER tablet (SRR). Test 6 (T6): 1 capsule BI 894416 Formulation F2, ER capsule (SRR).
  Interventions: Drug: BI 894416 Reference Formulation; Drug: BI 894416 Formulation A2; Drug: BI 894416 Formulation C2; Drug: BI 894416 Formulation D2; Drug: BI 894416 Formulation F2
- T2-T1-T3-R1-T4-T6 (sequence II+T6) (Experimental): Sequence II+T6, with treatments in the following order: T2-T1-T3-R1-T4-T6 with a washout period of at least 4 days between treatments. All test treatments (T1-T6) were one single dose of 62.5 milligram. R1 and T1-T4: taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. T5-T6: taken orally with 240 mL of water following a high-fat high-calorie breakfast.
  Reference (R1): 60 milligram (mg) (6 x 10 mg tablets) BI 894416 Reference Formulation, immediate release (IR) tablets.
  Test 1 (T1): 1 tablet BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR).
  Test 2 (T2): 1 tablet BI 894416 Formulation C2, ER tablet (slow release rate, SRR).
  Test 3 (T3): 1 capsule BI 894416 Formulation D2, ER capsule (FRR). Test 4 (T4): 1 capsule BI 894416 Formulation F2, ER capsule (SRR). Test 5 (T5): 1 tablet BI 894416 Formulation C2, ER tablet (SRR). Test 6 (T6): 1 capsule BI 894416 Formulation F2, ER capsule (SRR).
  Interventions: Drug: BI 894416 Reference Formulation; Drug: BI 894416 Formulation A2; Drug: BI 894416 Formulation C2; Drug: BI 894416 Formulation D2; Drug: BI 894416 Formulation F2
- T4-T3-R1-T2-T1-T5 (sequence III+T5) (Experimental): Sequence III+T5, with treatments in the following order: T4-T3-R1-T2-T1-T5 with a washout period of at least 4 days between treatments. All test treatments (T1-T6) were one single dose of 62.5 milligram. R1 and T1-T4: taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. T5-T6: taken orally with 240 mL of water following a high-fat high-calorie breakfast.
  Reference (R1): 60 milligram (mg) (6 x 10 mg tablets) BI 894416 Reference Formulation, immediate release (IR) tablets.
  Test 1 (T1): 1 tablet BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR).
  Test 2 (T2): 1 tablet BI 894416 Formulation C2, ER tablet (slow release rate, SRR).
  Test 3 (T3): 1 capsule BI 894416 Formulation D2, ER capsule (FRR). Test 4 (T4): 1 capsule BI 894416 Formulation F2, ER capsule (SRR). Test 5 (T5): 1 tablet BI 894416 Formulation C2, ER tablet (SRR). Test 6 (T6): 1 capsule BI 894416 Formulation F2, ER capsule (SRR).
  Interventions: Drug: BI 894416 Reference Formulation; Drug: BI 894416 Formulation A2; Drug: BI 894416 Formulation C2; Drug: BI 894416 Formulation D2; Drug: BI 894416 Formulation F2
- T4-T3-R1-T2-T1-T6 (sequence III+T6) (Experimental): Sequence III+T6, with treatments in the following order: T4-T3-R1-T2-T1-T6 with a washout period of at least 4 days between treatments. All test treatments (T1-T6) were one single dose of 62.5 milligram. R1 and T1-T4: taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. T5-T6: taken orally with 240 mL of water following a high-fat high-calorie breakfast.
  Reference (R1): 60 milligram (mg) (6 x 10 mg tablets) BI 894416 Reference Formulation, immediate release (IR) tablets.
  Test 1 (T1): 1 tablet BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR).
  Test 2 (T2): 1 tablet BI 894416 Formulation C2, ER tablet (slow release rate, SRR).
  Test 3 (T3): 1 capsule BI 894416 Formulation D2, ER capsule (FRR). Test 4 (T4): 1 capsule BI 894416 Formulation F2, ER capsule (SRR). Test 5 (T5): 1 tablet BI 894416 Formulation C2, ER tablet (SRR). Test 6 (T6): 1 capsule BI 894416 Formulation F2, ER capsule (SRR).
  Interventions: Drug: BI 894416 Reference Formulation; Drug: BI 894416 Formulation A2; Drug: BI 894416 Formulation C2; Drug: BI 894416 Formulation D2; Drug: BI 894416 Formulation F2
- T1-T4-T2-T3-R1-T5 (sequence IV+T5) (Experimental): Sequence IV+T5, with treatments in the following order: T1-T4-T2-T3-R1-T5 with a washout period of at least 4 days between treatments. All test treatments (T1-T6) were one single dose of 62.5 milligram. R1 and T1-T4: taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. T5-T6: taken orally with 240 mL of water following a high-fat high-calorie breakfast.
  Reference (R1): 60 milligram (mg) (6 x 10 mg tablets) BI 894416 Reference Formulation, immediate release (IR) tablets.
  Test 1 (T1): 1 tablet BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR).
  Test 2 (T2): 1 tablet BI 894416 Formulation C2, ER tablet (slow release rate, SRR).
  Test 3 (T3): 1 capsule BI 894416 Formulation D2, ER capsule (FRR). Test 4 (T4): 1 capsule BI 894416 Formulation F2, ER capsule (SRR). Test 5 (T5): 1 tablet BI 894416 Formulation C2, ER tablet (SRR). Test 6 (T6): 1 capsule BI 894416 Formulation F2, ER capsule (SRR).
  Interventions: Drug: BI 894416 Reference Formulation; Drug: BI 894416 Formulation A2; Drug: BI 894416 Formulation C2; Drug: BI 894416 Formulation D2; Drug: BI 894416 Formulation F2
- T1-T4-T2-T3-R1-T6 (sequence IV+T6) (Experimental): Sequence IV+T6, with treatments in the following order: T1-T4-T2-T3-R1-T6 with a washout period of at least 4 days between treatments. All test treatments (T1-T6) were one single dose of 62.5 milligram. R1 and T1-T4: taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. T5-T6: taken orally with 240 mL of water following a high-fat high-calorie breakfast.
  Reference (R1): 60 milligram (mg) (6 x 10 mg tablets) BI 894416 Reference Formulation, immediate release (IR) tablets.
  Test 1 (T1): 1 tablet BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR).
  Test 2 (T2): 1 tablet BI 894416 Formulation C2, ER tablet (slow release rate, SRR).
  Test 3 (T3): 1 capsule BI 894416 Formulation D2, ER capsule (FRR). Test 4 (T4): 1 capsule BI 894416 Formulation F2, ER capsule (SRR). Test 5 (T5): 1 tablet BI 894416 Formulation C2, ER tablet (SRR). Test 6 (T6): 1 capsule BI 894416 Formulation F2, ER capsule (SRR).
  Interventions: Drug: BI 894416 Reference Formulation; Drug: BI 894416 Formulation A2; Drug: BI 894416 Formulation C2; Drug: BI 894416 Formulation D2; Drug: BI 894416 Formulation F2
- R1-T2-T4-T1-T3-T5 (sequence V+T5) (Experimental): Sequence V+T5, with treatments in the following order: R1-T2-T4-T1-T3-T5 with a washout period of at least 4 days between treatments. All test treatments (T1-T6) were one single dose of 62.5 milligram. R1 and T1-T4: taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. T5-T6: taken orally with 240 mL of water following a high-fat high-calorie breakfast.
  Reference (R1): 60 milligram (mg) (6 x 10 mg tablets) BI 894416 Reference Formulation, immediate release (IR) tablets.
  Test 1 (T1): 1 tablet BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR).
  Test 2 (T2): 1 tablet BI 894416 Formulation C2, ER tablet (slow release rate, SRR).
  Test 3 (T3): 1 capsule BI 894416 Formulation D2, ER capsule (FRR). Test 4 (T4): 1 capsule BI 894416 Formulation F2, ER capsule (SRR). Test 5 (T5): 1 tablet BI 894416 Formulation C2, ER tablet (SRR). Test 6 (T6): 1 capsule BI 894416 Formulation F2, ER capsule (SRR).
  Interventions: Drug: BI 894416 Reference Formulation; Drug: BI 894416 Formulation A2; Drug: BI 894416 Formulation C2; Drug: BI 894416 Formulation D2; Drug: BI 894416 Formulation F2
- R1-T2-T4-T1-T3-T6 (sequence V+T6) (Experimental): Sequence V+T6, with treatments in the following order: R1-T2-T4-T1-T3-T6with a washout period of at least 4 days between treatments. All test treatments (T1-T6) were one single dose of 62.5 milligram. R1 and T1-T4: taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. T5-T6: taken orally with 240 mL of water following a high-fat high-calorie breakfast.
  Reference (R1): 60 milligram (mg) (6 x 10 mg tablets) BI 894416 Reference Formulation, immediate release (IR) tablets.
  Test 1 (T1): 1 tablet BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR).
  Test 2 (T2): 1 tablet BI 894416 Formulation C2, ER tablet (slow release rate, SRR).
  Test 3 (T3): 1 capsule BI 894416 Formulation D2, ER capsule (FRR). Test 4 (T4): 1 capsule BI 894416 Formulation F2, ER capsule (SRR). Test 5 (T5): 1 tablet BI 894416 Formulation C2, ER tablet (SRR). Test 6 (T6): 1 capsule BI 894416 Formulation F2, ER capsule (SRR).
  Interventions: Drug: BI 894416 Reference Formulation; Drug: BI 894416 Formulation A2; Drug: BI 894416 Formulation C2; Drug: BI 894416 Formulation D2; Drug: BI 894416 Formulation F2

INTERVENTIONS:
Drug: BI 894416 Reference Formulation — R1 - 60 milligram (6 x 10 milligram tablets) BI 894416 Reference Formulation, immediate release (IR) tablets taken orally with 240 mL of water after an overnight fast of at least 10 hours.
Drug: BI 894416 Formulation A2 — T1 - One single dose of 62.5 milligram (1 tablet) BI 894416 Formulation A2, extended release (ER) tablet (fast release rate, FRR) taken orally with 240 mL of water after an overnight fast of at least 10 hours.
Drug: BI 894416 Formulation C2 — T2 - One single dose of 62.5 milligram (1 tablet) BI 894416 Formulation C2, extended release (ER) tablet (slow release rate, SRR) taken orally with 240 mL of water after an overnight fast of at least 10 hours.
  and T5 - One single dose of 62.5 milligram (1 tablet) BI 894416 Formulation C2, extended release (ER) tablet (slow release rate, SRR) taken orally with 240 mL of water following a high-fat high-calorie breakfast.
Drug: BI 894416 Formulation D2 — T3 - One single dose of 62.5 milligram (1 capsule) BI 894416 Formulation D2, extended release (ER) capsule (fast release rate, FRR) taken orally with 240 mL of water after an overnight fast of at least 10 hours.
Drug: BI 894416 Formulation F2 — T4 - One single dose of 62.5 milligram (1 capsule) BI 894416 Formulation F2, extended release (ER) capsule (slow release rate, SRR) taken orally with 240 mL of water after an overnight fast of at least 10 hours.
  and T6 - One single dose of 62.5 milligram (1 capsule) BI 894416 Formulation F2, extended release (ER) capsule (slow release rate, SRR) taken orally with 240 mL of water following a high-fat high-calorie breakfast.

SUMMARY:
The main objective of this trial is to select a formulation principle (tablet vs. capsule) and to optimize the identified extended release formulation of BI 894416, if needed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive) at the time of signing informed consent
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive) as measured at screening
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Subjects who are sexually active must use, with their partner, highly effective contraception from the time of administration of trial medication until 30 days after administration of trial medication. Adequate methods are:

  * Condoms plus use of hormonal contraception by the female partner that started at least 2 months prior to administration of trial medication (e.g., implants, injectables, combined oral or vaginal contraceptives, intrauterine device) or
  * Condoms plus surgical sterilization (vasectomy at least 1 year prior to enrolment) or
  * Condoms plus surgically sterilised partner (including hysterectomy) or
  * Condoms plus intrauterine device or
  * Condoms plus partner of non-childbearing potential (including homosexual men) Subjects are required to use condoms to prevent unintended exposure of the partner (both, male and female) to the study drug via seminal fluid. Male subjects should use a condom throughout the study and for 30 days after last Investigational Medicinal Product (IMP) administration. Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, with their partner, they must comply with the contraceptive requirements detailed above Male subjects should not donate sperm for the duration of the study and for at least 30 days after last IMP administration

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR), Electrocardiogram (ECG), physical and neurological examination) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 40 to 90 mmHg, or pulse rate outside the range of 40 to 100 bpm at screening and pre-dose of first period
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients). Inactive hayfever is permitted.
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 90 days of planned first administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (unless the subject quit smoking for at least 3 months prior to first planned administration of trial medication) as demonstrated by a positive urine cotinine test; this includes also the use of e-cigarettes and nicotine replacement products
* Alcohol abuse (consumption of more than 21 units per week) or positive alcohol breath test
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening and predose
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* History of relevant neurological disorder affecting the peripheral or central nervous system (this includes but is not limited to: stroke, epilepsy, inflammatory or atrophic diseases affecting the nervous system, cluster headache or any cancer of the nervous system). Febrile seizures in childhood or adolescence, recovered carpal tunnel syndrome, recovered uncomplicated meningitis, recovered herpes zoster, tension headache, occasional benign tics (e.g. due to stress) or minor par- or dysesthesia (e.g. as a side effect of prior blood withdrawal) do not constitute a history of relevant neurological disorder.
* History of immunological disease, except allergy not relevant to the trial (such as mild hay fever or dust mite allergy) and except asthma in childhood or adolescence
* History of cancer (other than successfully treated basal cell carcinoma)
* Liver enzymes (ALT, AST, GGT, AP) above upper limit of normal at the screening examination
* Within 10 days prior to administration of trial medication, use of any drug that could reasonably inhibit platelet aggregation or coagulation (e.g., acetylsalicylic acid)
* Male subjects with Woman of child bearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of first administration of trial medication until 30 days after the last administration of trial medication
* Subjects with pregnant or lactating partners

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Formulation selection and subsequent optimization of two different oral formulations of BI 894416 in healthy male subjects (open-label, randomised, single-dose study in two parts; trial part 1: five-period crossover design with an additional sixth period in a fixed sequence; (optional) trial part 2: three-period crossover followed by a two-period crossover design), trial part 2 was not performed.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Treatment Period 1 + Washout
Arm/Group | T3-R1-T1-T4-T2-T5 (Sequence I+T5) | T3-R1-T1-T4-T2-T6 (Sequence I+T6) | T2-T1-T3-R1-T4-T5 (Sequence II+T5) | T2-T1-T3-R1-T4-T6 (Sequence II+T6) | T4-T3-R1-T2-T1-T5 (Sequence III+T5) | T4-T3-R1-T2-T1-T6 (Sequence III+T6) | T1-T4-T2-T3-R1-T5 (Sequence IV+T5) | T1-T4-T2-T3-R1-T6 (Sequence IV+T6) | R1-T2-T4-T1-T3-T5 (Sequence V+T5) | R1-T2-T4-T1-T3-T6 (Sequence V+T6)
Started | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Completed | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 + Washout
Arm/Group | T3-R1-T1-T4-T2-T5 (Sequence I+T5) | T3-R1-T1-T4-T2-T6 (Sequence I+T6) | T2-T1-T3-R1-T4-T5 (Sequence II+T5) | T2-T1-T3-R1-T4-T6 (Sequence II+T6) | T4-T3-R1-T2-T1-T5 (Sequence III+T5) | T4-T3-R1-T2-T1-T6 (Sequence III+T6) | T1-T4-T2-T3-R1-T5 (Sequence IV+T5) | T1-T4-T2-T3-R1-T6 (Sequence IV+T6) | R1-T2-T4-T1-T3-T5 (Sequence V+T5) | R1-T2-T4-T1-T3-T6 (Sequence V+T6)
Started | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Completed | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 + Washout
Arm/Group | T3-R1-T1-T4-T2-T5 (Sequence I+T5) | T3-R1-T1-T4-T2-T6 (Sequence I+T6) | T2-T1-T3-R1-T4-T5 (Sequence II+T5) | T2-T1-T3-R1-T4-T6 (Sequence II+T6) | T4-T3-R1-T2-T1-T5 (Sequence III+T5) | T4-T3-R1-T2-T1-T6 (Sequence III+T6) | T1-T4-T2-T3-R1-T5 (Sequence IV+T5) | T1-T4-T2-T3-R1-T6 (Sequence IV+T6) | R1-T2-T4-T1-T3-T5 (Sequence V+T5) | R1-T2-T4-T1-T3-T6 (Sequence V+T6)
Started | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Completed | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4 + Washout
Arm/Group | T3-R1-T1-T4-T2-T5 (Sequence I+T5) | T3-R1-T1-T4-T2-T6 (Sequence I+T6) | T2-T1-T3-R1-T4-T5 (Sequence II+T5) | T2-T1-T3-R1-T4-T6 (Sequence II+T6) | T4-T3-R1-T2-T1-T5 (Sequence III+T5) | T4-T3-R1-T2-T1-T6 (Sequence III+T6) | T1-T4-T2-T3-R1-T5 (Sequence IV+T5) | T1-T4-T2-T3-R1-T6 (Sequence IV+T6) | R1-T2-T4-T1-T3-T5 (Sequence V+T5) | R1-T2-T4-T1-T3-T6 (Sequence V+T6)
Started | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Completed | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 5 + Washout
Arm/Group | T3-R1-T1-T4-T2-T5 (Sequence I+T5) | T3-R1-T1-T4-T2-T6 (Sequence I+T6) | T2-T1-T3-R1-T4-T5 (Sequence II+T5) | T2-T1-T3-R1-T4-T6 (Sequence II+T6) | T4-T3-R1-T2-T1-T5 (Sequence III+T5) | T4-T3-R1-T2-T1-T6 (Sequence III+T6) | T1-T4-T2-T3-R1-T5 (Sequence IV+T5) | T1-T4-T2-T3-R1-T6 (Sequence IV+T6) | R1-T2-T4-T1-T3-T5 (Sequence V+T5) | R1-T2-T4-T1-T3-T6 (Sequence V+T6)
Started | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Completed | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 6
Arm/Group | T3-R1-T1-T4-T2-T5 (Sequence I+T5) | T3-R1-T1-T4-T2-T6 (Sequence I+T6) | T2-T1-T3-R1-T4-T5 (Sequence II+T5) | T2-T1-T3-R1-T4-T6 (Sequence II+T6) | T4-T3-R1-T2-T1-T5 (Sequence III+T5) | T4-T3-R1-T2-T1-T6 (Sequence III+T6) | T1-T4-T2-T3-R1-T5 (Sequence IV+T5) | T1-T4-T2-T3-R1-T6 (Sequence IV+T6) | R1-T2-T4-T1-T3-T5 (Sequence V+T5) | R1-T2-T4-T1-T3-T6 (Sequence V+T6)
Started | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Completed | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This analysis set included all subjects who were randomised and received at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | T3-R1-T1-T4-T2-T5 (Sequence I+T5) | T3-R1-T1-T4-T2-T6 (Sequence I+T6) | T2-T1-T3-R1-T4-T5 (Sequence II+T5) | T2-T1-T3-R1-T4-T6 (Sequence II+T6) | T4-T3-R1-T2-T1-T5 (Sequence III+T5) | T4-T3-R1-T2-T1-T6 (Sequence III+T6) | T1-T4-T2-T3-R1-T5 (Sequence IV+T5) | T1-T4-T2-T3-R1-T6 (Sequence IV+T6) | R1-T2-T4-T1-T3-T5 (Sequence V+T5) | R1-T2-T4-T1-T3-T6 (Sequence V+T6) | Total
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (17.7) | 37.0 (0.0) | 29.5 (7.8) | 30.3 (4.0) | 39.0 (8.5) | 31.5 (2.1) | 30.0 (8.2) | 43.3 (13.2) | 25.0 (4.2) | 25.3 (5.9) | 32.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 3 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: Within 3 hours before and 0.33, 0.66, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24, 34, 48, 58 and 72 hours following drug administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This analysis set included all subjects who were randomised, received at least one dose of trial medication and who provided at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomol/Liter
Groups:
- Reference 1 - BI 894416 Reference Formulation Tablet, Fasted: 60 milligram (6 x 10 milligram tablets) BI 894416 Reference Formulation, immediate release (IR) tablets taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours.
- Test 1 - BI 894416 Fast Release Rate (FRR) Tablet, Fasted: One single tablet of 62.5 milligram BI 894416 Formulation A2, extended release (ER) tablet (fast release rate (FRR)) taken orally with 240 mL of water after an overnight fast of at least 10 hours.
- Test 2 - BI 894416 Slow Release Rate (SRR) Tablet, Fasted: One single tablet of 62.5 milligram BI 894416 Formulation C2, ER tablet (slow release rate (SRR)) taken orally with 240 mL of water after an overnight fast of at least 10 hours.
- Test 3 - BI 894416 Fast Release Rate (FRR) Capsule, Fasted: One single capsule of 62.5 milligram BI 894416 Formulation D2, ER capsule (FRR) taken orally with 240 mL of water after an overnight fast of at least 10 hours.
- Test 4 - BI 894416 Slow Release Rate (SRR) Capsule, Fasted: One single capsule of 62.5 milligram BI 894416 Formulation F2, ER capsule (SRR) taken orally with 240 mL of water after an overnight fast of at least 10 hours.
- Test 5 - BI 894416 Slow Release Rate (SRR) Tablet, Fed: One single tablet of 62.5 milligram BI 894416 Formulation C2, ER tablet (SRR) taken orally with 240 mL of water following a high-fat high-calorie breakfast.
- Test 6 - BI 894416 Slow Release Rate (SRR) Capsule, Fed: One single capsule of 62.5 milligram BI 894416 Formulation F2, ER capsule (SRR) taken orally with 240 mL of water following a high-fat high-calorie breakfast.
Arm/Group | Reference 1 - BI 894416 Reference Formulation Tablet, Fasted | Test 1 - BI 894416 Fast Release Rate (FRR) Tablet, Fasted | Test 2 - BI 894416 Slow Release Rate (SRR) Tablet, Fasted | Test 3 - BI 894416 Fast Release Rate (FRR) Capsule, Fasted | Test 4 - BI 894416 Slow Release Rate (SRR) Capsule, Fasted | Test 5 - BI 894416 Slow Release Rate (SRR) Tablet, Fed | Test 6 - BI 894416 Slow Release Rate (SRR) Capsule, Fed
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 11 | 13
hour*nanomol/Liter | 9800 (30.6) | 8260 (29.6) | 7030 (31.7) | 9100 (33.3) | 7430 (35.8) | 9680 (31.1) | 8930 (24.8)
Statistical Analysis 1: Comparison: Reference 1 - BI 894416 Reference Formulation Tablet, Fasted vs Test 1 - BI 894416 Fast Release Rate (FRR) Tablet, Fasted; Analysis of variance (ANOVA) model on the logarithmic scale, including effects accounting for 'sequence', 'subjects nested within sequences', 'period', and 'treatment' (formulation). The effect 'subjects within sequences' was to be considered as random, while the other effects were to be considered as fixed; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 85.9, 90% CI 2-sided [80.3 to 91.7] — Test/reference, intra-individual geometric coefficient of variance (gCV) =13.9
Statistical Analysis 2: Comparison: Reference 1 - BI 894416 Reference Formulation Tablet, Fasted vs Test 2 - BI 894416 Slow Release Rate (SRR) Tablet, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 72.6, 90% CI 2-sided [68.0 to 77.6] — Test/reference, intra-individual geometric coefficient of variance (gCV) =13.9
Statistical Analysis 3: Comparison: Reference 1 - BI 894416 Reference Formulation Tablet, Fasted vs Test 3 - BI 894416 Fast Release Rate (FRR) Capsule, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 92.4, 90% CI 2-sided [86.5 to 98.8] — Test/reference, intra-individual geometric coefficient of variance (gCV) =13.9
Statistical Analysis 4: Comparison: Reference 1 - BI 894416 Reference Formulation Tablet, Fasted vs Test 4 - BI 894416 Slow Release Rate (SRR) Capsule, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 76.6, 90% CI 2-sided [71.6 to 81.8] — Test/reference, intra-individual geometric coefficient of variance (gCV) =13.9
Statistical Analysis 5: Comparison: Test 2 - BI 894416 Slow Release Rate (SRR) Tablet, Fasted vs Test 5 - BI 894416 Slow Release Rate (SRR) Tablet, Fed; Analysis of variance (ANOVA) model on the logarithmic scale, including effects accounting for 'subjects' and 'treatment'. The effect 'subjects' were to be considered as random, while the effect 'treatment' was to be considered as fixed; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 133.4, 90% CI 2-sided [117.2 to 151.9] — Test/reference, intra-individual geometric coefficient of variance (gCV) =17.6
Statistical Analysis 6: Comparison: Test 4 - BI 894416 Slow Release Rate (SRR) Capsule, Fasted vs Test 6 - BI 894416 Slow Release Rate (SRR) Capsule, Fed; [analysis description as in outcome 1, analysis 5]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 114.2, 90% CI 2-sided [102.3 to 127.6] — Test/reference, intra-individual geometric coefficient of variance (gCV) =16.2

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomol/Liter
Arm/Group | Reference 1 - BI 894416 Reference Formulation Tablet, Fasted | Test 1 - BI 894416 Fast Release Rate (FRR) Tablet, Fasted | Test 2 - BI 894416 Slow Release Rate (SRR) Tablet, Fasted | Test 3 - BI 894416 Fast Release Rate (FRR) Capsule, Fasted | Test 4 - BI 894416 Slow Release Rate (SRR) Capsule, Fasted | Test 5 - BI 894416 Slow Release Rate (SRR) Tablet, Fed | Test 6 - BI 894416 Slow Release Rate (SRR) Capsule, Fed
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 11 | 13
hour*nanomol/Liter | 9780 (30.5) | 8200 (29.5) | 6950 (31.8) | 9050 (33.2) | 7310 (36.3) | 9600 (30.6) | 8850 (24.9)
Statistical Analysis 1: Comparison: Reference 1 - BI 894416 Reference Formulation Tablet, Fasted vs Test 1 - BI 894416 Fast Release Rate (FRR) Tablet, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 85.5, 90% CI 2-sided [80.0 to 91.4] — Test/reference, intra-individual geometric coefficient of variance (gCV) =14.0
Statistical Analysis 2: Comparison: Reference 1 - BI 894416 Reference Formulation Tablet, Fasted vs Test 2 - BI 894416 Slow Release Rate (SRR) Tablet, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 72.1, 90% CI 2-sided [67.4 to 77.1] — Test/reference, intra-individual geometric coefficient of variance (gCV) =14.0
Statistical Analysis 3: Comparison: Reference 1 - BI 894416 Reference Formulation Tablet, Fasted vs Test 3 - BI 894416 Fast Release Rate (FRR) Capsule, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 92.2, 90% CI 2-sided [86.3 to 98.6] — Test/reference, intra-individual geometric coefficient of variance (gCV) =14.0
Statistical Analysis 4: Comparison: Reference 1 - BI 894416 Reference Formulation Tablet, Fasted vs Test 4 - BI 894416 Slow Release Rate (SRR) Capsule, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 75.5, 90% CI 2-sided [70.6 to 80.7] — Test/reference, intra-individual geometric coefficient of variance (gCV) =14.0
Statistical Analysis 5: Comparison: Test 2 - BI 894416 Slow Release Rate (SRR) Tablet, Fasted vs Test 5 - BI 894416 Slow Release Rate (SRR) Tablet, Fed; [analysis description as in outcome 1, analysis 5]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 134.2, 90% CI 2-sided [117.6 to 153.0] — Test/reference, intra-individual geometric coefficient of variance (gCV) =17.9
Statistical Analysis 6: Comparison: Test 4 - BI 894416 Slow Release Rate (SRR) Capsule, Fasted vs Test 6 - BI 894416 Slow Release Rate (SRR) Capsule, Fed; [analysis description as in outcome 1, analysis 5]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 114.8, 90% CI 2-sided [102.9 to 128.1] — Test/reference, intra-individual geometric coefficient of variance (gCV) =16.1

ADVERSE EVENTS:
Time Frame: From the first administration of BI 894416 in any formulation until the subject's trial termination date, up to days 35 days.
Description: Treated set (TS): This analysis set included all subjects who were randomised and received at least one dose of trial medication.
  In accordance with the protocol, all study arms used the same active substance (BI 894416) in the same dosage and were combined for safety reporting as no safety issues were expected with any specific formulation.
Arm/Group | Reference 1 - BI 894416 Reference Formulation Tablet, Fasted | Test 1 - BI 894416 Fast Release Rate (FRR) Tablet, Fasted | Test 2 - BI 894416 Slow Release Rate (SRR) Tablet, Fasted | Test 3 - BI 894416 Fast Release Rate (FRR) Capsule, Fasted | Test 4 - BI 894416 Slow Release Rate (SRR) Capsule, Fasted | Test 5 - BI 894416 Slow Release Rate (SRR) Tablet, Fed | Test 6 - BI 894416 Slow Release Rate (SRR) Capsule, Fed
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 1/24 | 1/24 | 3/24 | 2/24 | 2/24 | 3/11 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reference 1 - BI 894416 Reference Formulation Tablet, Fasted (N=24) | Test 1 - BI 894416 Fast Release Rate (FRR) Tablet, Fasted (N=24) | Test 2 - BI 894416 Slow Release Rate (SRR) Tablet, Fasted (N=24) | Test 3 - BI 894416 Fast Release Rate (FRR) Capsule, Fasted (N=24) | Test 4 - BI 894416 Slow Release Rate (SRR) Capsule, Fasted (N=24) | Test 5 - BI 894416 Slow Release Rate (SRR) Tablet, Fed (N=11) | Test 6 - BI 894416 Slow Release Rate (SRR) Capsule, Fed (N=13)
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT04232839/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT04232839/SAP_001.pdf